CLINICAL TRIAL: NCT01314118
Title: A Multicenter, Open-label, Single-arm, Phase 2 Study of Abiraterone Acetate Plus Prednisone in Subjects With Advanced Prostate Cancer Without Radiographic Evidence of Metastatic Disease
Brief Title: IMAAGEN: Impact of Abiraterone Acetate in Prostate-Specific Antigen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017932; 212082PCR2005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-03-04; First posted 2011-03-14 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Prostatic Neoplasm
Keywords: abiraterone acetate; prednisone; zytiga
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 001 (Experimental): abiraterone acetate in combination with prednisone Abiraterone acetate will be taken as 4 x 250 mg tablets by mouth (PO) once daily. Prednisone will be taken as 2 x 2.5 mg tablets PO once daily.
  Interventions: Drug: abiraterone acetate in combination with prednisone

INTERVENTIONS:
Drug: abiraterone acetate in combination with prednisone — Abiraterone acetate will be taken as 4 x 250 mg tablets by mouth (PO) once daily. Prednisone will be taken as 2 x 2.5 mg tablets PO once daily.

SUMMARY:
The purpose of this study is to show that abiraterone acetate plus prednisone added to the current standard of care, gonadotropin-releasing hormone (GnRH) decreases prostate specific antigen (PSA) and prolongs the time until it is evident that the cancer has grown. Additionally, safety information about abiraterone acetate in combination with prednisone will be collected. This will include looking at what side effects occur, how often they occur, and for how long they last.

DETAILED DESCRIPTION:
This is a Phase 2, prospective, multicenter, open-label, single-arm study of abiraterone acetate plus prednisone in men with non-metastatic, castration-resistant prostate cancer (CRPC) who have a rising PSA despite castrate levels of testosterone. The study consists of Screening Phase (up to 4 weeks), Core Study Treatment Phase (comprised of six 28-day cycles), a Pre-metastatic Disease Follow-up Phase, an Optional Drug Holiday Phase; and a 30-day Safety Follow-up Visit. Each treatment cycle will last 28 days. Participating participants will receive study agents (Abiraterone acetate 1000 mg/day plus prednisone 5 mg/day, orally) continually during the study. If the partcipants elects to participate in the Optional Drug Holiday Phase, participants will discontinue abiraterone acetate plus prednisone and ADT. Participants will have the option to return to study medication during the first year of the Optional Drug Holiday Phase if there is evidence of rising PSA but no metastasis based on study imaging. If participants do no elect to participate, they will continue with the core study treatment as per protocol. The study will end when all participated participants have disease progression or end of the 2-year period (if participants participated in the Optional Drug Holiday Phase). Participants will be required to return to the study site 30 days after receiving the last dose of abiraterone acetate for safety follow-up.

ELIGIBILITY:
Major Inclusion Criteria:

* Be a male >= 18 years of age
* Have adenocarcinoma of the prostate
* Currently receiving continuous treatment with Gonadotropin-releasing hormone (GnRH) monotherapy for at least 6 months before or have undergone surgical removal of the testicles
* Serum testosterone of < 50 ng/dL(< 2.0 nM)
* Have rising PSA defined as a PSA of >= 10 ng/mL obtained at screening or PSADT of ≤ 10 months with the first of the 3 consecutive PSA values used to calculate PSADT ≥ 2.0 ng/mL
* Have an Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Be capable of swallowing study agents whole as a tablet
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol

Major Exclusion Criteria:

* Have prior or current evidence of local disease progression or metastatic disease as defined by modified response evaluation criteria in solid tumors (RECIST) criteria
* Have received chemotherapy for treatment of castrate-resistant prostate cancer; however, if a patient received chemotherapy in an adjuvant setting, prior to having CRPC, for castrate-sensitive prostate cancer, the patient is still eligible
* Are currently receiving any antiandrogen therapy (eg, bicalutamide, flutamide, or nilutamide).
* If previously treated with antiandrogen therapy, there must be documentation of at least 2 consecutive rising PSA values at least 2 weeks apart obtained prior to screening
* If previously treated with flutamide, at least 1 of the PSA values must be obtained 4 weeks or more after flutamide discontinuation.
* If previously treated with bicalutamide or nilutamide, at least 1 of the PSA values must be obtained 6 weeks or more after antiandrogen discontinuation
* Have previously received agents having any CYP17 inhibitory activity for the treatment of prostate cancer, such as ketoconazole
* Have previously received aminoglutethimide
* Have an active infection or other medical condition that would contraindicate prednisone use
* Have uncontrolled hypertension
* Have active hepatitis or chronic liver disease
* Have clinically significant heart disease
* Have poorly controlled diabetes
* Have received an investigational therapeutic within 30 days of screening
* Have partners of childbearing potential and are not willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 1 week after last dose of abiraterone acetate.
* Individuals with a history of a non-prostate malignancy are ineligible for this study with the following exceptions. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: basal cell or squamous cell carcinoma of the skin

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-05-04 (Actual); Primary Completion 2013-12-24 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Services, LLC. Clinical Trial, Study Director — Janssen Biotech, Inc.
Locations (45):
- United States (45):
  - Homewood, Alabama
  - Huntsville, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Denver, Colorado
  - Aventura, Florida
  - Orange City, Florida
  - Atlanta, Georgia
  - Evanston, Illinois
  - Galesburg, Illinois
  - Glenview, Illinois
  - Melrose Park, Illinois
  - Fort Wayne, Indiana
  - Jeffersonville, Indiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Lansing, Michigan
  - Omaha, Nebraska
  - Lawrenceville, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - Buffalo, New York
  - Garden City, New York
  - New York, New York
  - Poughkeepsie, New York
  - Staten Island, New York
  - Chapel Hill, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate Plus Prednisone: Participants were given abiraterone acetate 1000 milligrams (mg) (4*250 mg) tablets plus prednisone 5 mg (2*2.5 mg) tablets orally once daily in core study treatment phase (comprised of 6, 28-day cycles). After the core study treatment phase, participants who entered the pre-metastatic disease follow-up phase continued the study treatment until radiographic confirmation of disease progression, intolerable toxicity, investigator's decision, and withdrawal by participant or until the sponsor decided to stop the trial. As per amendment 6, participants who opted for the drug holiday phase stopped abiraterone acetate plus prednisone, and androgen-deprivation therapy (ADT), with the option to restart treatment within the first year if prostate-specific antigen (PSA) levels increased without metastasis. Those who did not opt for the drug holiday phase continued treatment. The study ended when all participants had disease progression or completed the 2-year period (for drug holiday participants) (up to 140 months; 153 Cycles). Post-metastatic disease follow-up phase was also discontinued, though participants already enrolled at the time of protocol amendment 6 remained on study. A safety follow-up visit was required 30 days after the last dose of abiraterone acetate.
Period: Overall Study
Arm/Group | Abiraterone Acetate Plus Prednisone
Started | 131
Completed Until Treatment Cycle 6 | 112
Completed (Completed refers to patients at clinical cut-off with no evidence of disease progression who continued on treatment whereas Not Completed refers to patients who discontinued treatment.) | 47
Not Completed | 84
Not completed — Adverse Event | 10
Not completed — Progressive disease | 3
Not completed — Death | 8
Not completed — Physician Decision | 13
Not completed — Sponsor Decision | 1
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 26
Not completed — Other | 21

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.2 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 131
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 108
  More than one race | 0
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 122
  Unknown or Not Reported | 1
  Hispanic or Latino | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 131

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 50 Percent (%) Reduction in Prostate-Specific Antigen (PSA) During the Core Study
Description: Percentage of participants with greater than or equal to 50 percent decrease in PSA levels was assessed.
Time Frame: End of core study visit (Approximately at Month 6)
Population: Efficacy evaluable set included all participants who received at least one dose of study drug, completed at least 1 cycle of treatment and had at least 1 post-baseline PSA assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 122
Percentage of participants | 86.9 [80.9 to 92.9]

2. Secondary Outcome: Time to Radiographic Evidence of Disease Progression (TTRP)
Description: Time to radiographic evidence of disease progression is defined as the time interval from the date of enrollment (Day 1) to the date of disease progression. A participant was considered as progressed by bone scan if: 1) The appearance of greater than or equal to (>=) 2 new lesions, and, following the first assessment, a confirmatory scan performed 6 or more weeks later that shows a minimum of 2 or more additional new lesions, 2) If >=2 new lesions are seen on scans following the first assessment, the confirmation is still required after 6 weeks; however, 2 addition lesions are not required to confirm progression, and 3) The date of progression is the date of the first scan that shows the changes.
Time Frame: Maximum up to Month 30.5
Population: All enrolled set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 131
Months | 41.4 [27.6 to NA] — Data was not evaluable as insufficient number of participants had the event.

3. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: Time to PSA progression is defined as the time interval from the date of enrollment (Day 1) to the date of first evidence of PSA progression. A participant was considered to have a PSA progression if the PSA level had a 25 percent (%) or greater increase and an absolute increase of 2 nanogram (ng)/milliliter (mL) or more, which is confirmed by a second value obtained in 3 or more weeks.
Time Frame: Maximum up to Month 30.5
Population: All enrolled set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 131
Months | 28.7 [21.2 to 38.2]

4. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 50 Percent (%) Reduction in Prostate-Specific Antigen (PSA) Levels After 3 Cycles of Treatment
Description: Percentage of participants with greater than or equal to 50 percent decrease in PSA levels was assessed. Decrease in PSA levels represented improvement.
Time Frame: End of Cycle 3 (Approximately Month 3)
Population: Efficacy evaluable set included all participants who received at least 1 dose of study drug, completed at least 1 cycle of treatment and had at least 1 post-baseline PSA assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Abiraterone Acetate Plus Prednisone
Number analyzed (Participants) | 122
Percentage of Participants | 85.2 [79.0 to 91.5]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From screening (-28 days) up to 141 months; Serious and Other AEs: From Cycle 1 Day 1 up to 30 days after last dose (up to 141 months)
Description: Safety evaluable set defined as all participants exposed to study agents (Abiraterone acetate or Prednisone).
Arm/Group | Abiraterone Acetate Plus Prednisone
All-Cause Mortality (participants affected / at risk) | 11/131
Serious Adverse Events (participants affected / at risk) | 61/131
Other Adverse Events (participants affected / at risk) | 120/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate Plus Prednisone (N=131)
Anaemia (Blood and lymphatic system disorders) | 2
Acute Myocardial Infarction (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 2
Cardiac Failure (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 2
Cardio-Respiratory Arrest (Cardiac disorders) | 2
Coronary Artery Disease (Cardiac disorders) | 4
Myocardial Infarction (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Meniere's Disease (Ear and labyrinth disorders) | 1
Adrenal Mass (Endocrine disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Colitis Ulcerative (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Obstruction Gastric (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 2
Rectourethral Fistula (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 2
Oedema Peripheral (General disorders) | 1
Systemic Inflammatory Response Syndrome (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Chest Wall Abscess (Infections and infestations) | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1
Giardiasis (Infections and infestations) | 1
Lobar Pneumonia (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Postoperative Wound Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 7
Septic Shock (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 4
Urosepsis (Infections and infestations) | 5
Cystitis Radiation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 2
Hip Fracture (Injury, poisoning and procedural complications) | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Transplant Failure (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 4
Blood Glucose Increased (Investigations) | 1
Blood Potassium Increased (Investigations) | 1
Hepatic Enzyme Increased (Investigations) | 1
Liver Function Test Abnormal (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 3
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1
Failure to Thrive (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Lactic Acidosis (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance Disorder (Nervous system disorders) | 1
Brain Mass (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Neurological Symptom (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 5
Acute Psychosis (Psychiatric disorders) | 1
Bladder Obstruction (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 2
Obstructive Uropathy (Renal and urinary disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 2
Urinary Retention (Renal and urinary disorders) | 5
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Nephrectomy (Surgical and medical procedures) | 1
Transurethral Prostatectomy (Surgical and medical procedures) | 1
Arteriosclerosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypertensive Crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral Circulatory Failure (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate Plus Prednisone (N=131)
Anaemia (Blood and lymphatic system disorders) | 13
Cataract (Eye disorders) | 9
Constipation (Gastrointestinal disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 27
Dyspepsia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 21
Asthenia (General disorders) | 7
Chest Pain (General disorders) | 9
Fatigue (General disorders) | 56
Influenza Like Illness (General disorders) | 11
Oedema Peripheral (General disorders) | 34
Pyrexia (General disorders) | 7
Bronchitis (Infections and infestations) | 10
Influenza (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 18
Sinusitis (Infections and infestations) | 13
Upper Respiratory Tract Infection (Infections and infestations) | 22
Urinary Tract Infection (Infections and infestations) | 24
Contusion (Injury, poisoning and procedural complications) | 8
Fall (Injury, poisoning and procedural complications) | 16
Rib Fracture (Injury, poisoning and procedural complications) | 8
Alanine Aminotransferase Increased (Investigations) | 9
Aspartate Aminotransferase Increased (Investigations) | 9
Blood Creatine Phosphokinase Increased (Investigations) | 7
Blood Creatinine Increased (Investigations) | 8
Weight Decreased (Investigations) | 8
Decreased Appetite (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 13
Hypokalaemia (Metabolism and nutrition disorders) | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Back Pain (Musculoskeletal and connective tissue disorders) | 23
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 13
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Neck Pain (Musculoskeletal and connective tissue disorders) | 11
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 18
Dizziness (Nervous system disorders) | 27
Headache (Nervous system disorders) | 25
Paraesthesia (Nervous system disorders) | 8
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 10
Dysuria (Renal and urinary disorders) | 7
Haematuria (Renal and urinary disorders) | 21
Micturition Urgency (Renal and urinary disorders) | 10
Nocturia (Renal and urinary disorders) | 8
Pollakiuria (Renal and urinary disorders) | 13
Urinary Incontinence (Renal and urinary disorders) | 13
Urinary Retention (Renal and urinary disorders) | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 8
Hot Flush (Vascular disorders) | 14
Hypertension (Vascular disorders) | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days. The sponsor will not mandate modifications to scientific content and does not have the right to suppress information.

DOCUMENTS (2):
  • Study Protocol (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT01314118/Prot_000.pdf
  • Statistical Analysis Plan (2014-02-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT01314118/SAP_001.pdf